CLINICAL TRIAL: NCT01756534
Title: The Effectiveness of an Oxidized Cellulose Patch Hemostatic Agent in Thyroid Surgery: a Prospective Randomized Controlled Study
Brief Title: Oxidized Cellulose Hemostatic Agent in Thyroid Surgery: a Prospective Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-ZG-AA-0633-CTIL
Record Dates: First submitted 2012-12-19; First posted 2012-12-27 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Thyroid Nodule; Thyroid Diseases; Goiter
MeSH Terms: conditions — Thyroid Nodule; Thyroid Diseases; Goiter

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CONVENTIONAL HEMOSTASIS (No Intervention): patients for whom conventional surgical procedures (i. e., ligatures and bipolar electrocautery alone) were used to achieve hemostasis
- SURGICEL (Active Comparator): patients will receive an oxidized cellulose patch (Surgicel®) in addition to conventional surgical procedures (i. e., ligatures and bipolar electrocautery alone)
  Interventions: Device: SURGICEL

INTERVENTIONS:
Device: SURGICEL — Surgicel® (Johnson and Johnson, New Brunswick, NJ, USA), an oxidized cellulose hemostatic agent, is indicated in surgical procedures as an adjunct to hemostasis when control of bleeding by ligature or other conventional procedures is ineffective or impractical.
  Arms: SURGICEL

SUMMARY:
This single-blind prospective randomized study was designed to assess the efficacy and safety of the use of Surgicel® compared to the use of conventional surgical procedures (ligatures and bipolar electrocautery alone) to achieve hemostasis in thyroid surgery

DETAILED DESCRIPTION:
patients who require a thyroidectomy will be enrolled after informed consent will begiven. Prior to thyroidectomy, patients will be randomized to two groups: 1) use of conventional surgical procedures to achieve hemostasis,i.e., ligatures and bipolar electrocauterization alone, and 2) use of oxidized cellulose patch (Surgicel©) in addition to classical methods (ligature; bipolar electrocautery). All anticoagulants will be discontinued 10 days prior to the operation, if this will not be possible the patient will be excluded. The investigators will perform the specified procedure in accordance with accepted clinical practice standards. At the end of the thyroidectomy, a meticulous hemostasis will be achieved. Before wound closure, the sealed affiliation envelopes will be opened and 1-2×2 cm oxidized cellulose patch will be placed over the thyroid bed depending on patient randomization. Next, a suction drain will be placed. The drains will be removed when the secretion volume/day will be less than 20 cc.

All operations will be performed under general anesthesia by three head and neck surgeons who had experience in thyroid surgery. Outcome measures will include duration of operation, hemodynamic variables on emergence (blood pressure and heart rate), volume of secretion in the drain, time to removal of wound drain, length of postoperative hospital stay, and incidence of postoperative complications, i.e. hemorrhage, transient hypoparathyroidism, wound infection, seroma, and recurrent laryngeal nerve palsy. Evaluation of the postoperative course and recording of data will be done by one surgeons blinded to the intervention (MA). Follow-up for this study will be ended one month after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients who required a thyroidectomy

Exclusion Criteria:

* Unwilling or unable to consent
* Age < 18 years
* known allergy to oxidized cellulose
* Inability to discontinue use of anticoagulants 10 days before surgery
* Coagulopathy that could not be corrected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-03 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study was the postoperative volume of wound drainage | 1 WEEK

SECONDARY OUTCOMES:
The secondary endpoints were events of bleeding requiring wound exploration under anesthesia | 48 HOURS
duration of drain use | 1 WEEK

OTHER OUTCOMES:
hospitalization time | 1 WEEK

CONTACTS AND LOCATIONS:
Overall Officials: ZIV GIL, MD PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Quick MW, Naeve J, Davidson N, Lester HA. Incubation with horse serum increases viability and decreases background neurotransmitter uptake in Xenopus oocytes. Biotechniques. 1992 Sep;13(3):357-61. No abstract available. PMID 1356369
- [Background] Cotulbea S, Marin I, Golumba R, Barbos R, Epure V, Valean M, Anghel I. [Our clinical management in treating seromucous otitis]. Rev Chir Oncol Radiol O R L Oftalmol Stomatol Otorinolaringol. 1988 Oct-Dec;33(4):259-64. No abstract available. Romanian. PMID 2978438
- [Derived] Amit M, Binenbaum Y, Cohen JT, Gil Z. Effectiveness of an oxidized cellulose patch hemostatic agent in thyroid surgery: a prospective, randomized, controlled study. J Am Coll Surg. 2013 Aug;217(2):221-5. doi: 10.1016/j.jamcollsurg.2013.03.022. PMID 23870217